CLINICAL TRIAL: NCT05128344
Title: A Phase 3, Randomized, Open-Label Study to Evaluate the Efficacy and Safety of AMZ002, Compared to Vigabatrin, in the Treatment of Infantile Spasms
Brief Title: A Study to Evaluate Safety and Efficacy of AMZ002 Treatment, Compared With Vigabatrin in Participants With Infantile Spasms
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic decision
Sponsor: Amzell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMZ002-002; 2021-003015-26 (EudraCT Number)
Record Dates: First submitted 2021-11-09; First posted 2021-11-22 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Spasms, Infantile
Keywords: AMZ002; Vigabatrin; Seizures; Electroencephalograms; Infantile spasms; West syndrome; Central Nervous System Diseases; Epileptic Syndrome
MeSH Terms: conditions — Spasms, Infantile; Seizures; Central Nervous System Diseases; Epileptic Syndromes | interventions — Vigabatrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMZ002 (Experimental)
  Interventions: Drug: AMZ002 injectable solution, 0.5mg/mL
- Vigabatrin (Active Comparator)
  Interventions: Drug: Vigabatrin, oral

INTERVENTIONS:
Drug: AMZ002 injectable solution, 0.5mg/mL — Injectable solution
  Arms: AMZ002
Drug: Vigabatrin, oral — Oral administration
  Arms: Vigabatrin

SUMMARY:
The main purpose of this study is to evaluate the efficacy of AMZ002 compared to Vigabatrin in participants with newly diagnosed infantile spasms (IS).

ELIGIBILITY:
Inclusion Criteria:

* Participant has been diagnosed with IS within 6 weeks prior to Screening. Diagnostic criteria include both clinical spasms and an EEG pattern consistent with hypsarrhythmia or significant abnormality compatible with IS
* Participant has normal renal function as defined by an estimated glomerular filtration rate (eGFR) greater than [>] 60 milliliter/minute (mL/min)/1.73 m^2, calculated as eGFR = 0.413 × (height [Centimeter (cm)]/serum creatinine [milligrams per deciliter {mg/dL}])
* Participant's legally authorized representative (that is [i.e.], parent or guardian) must provide written informed consent obtained per Institutional Review Board (IRB) policy and requirements, consistent with the International Council for Harmonisation (ICH)
* Participant's parent/guardian is able to understand and willing to comply with study procedures and restrictions

Exclusion Criteria:

* Participant has been diagnosed with tuberous sclerosis
* Participant has acute illness considered clinically significant by the Investigator within 30 days prior to Screening
* Participant has a diagnosis of recent systemic fungal infection; history of ocular herpes simplex; history of or current peptic ulcer; uncontrolled hypertension or congestive heart failure; or any other condition that would be significantly impacted by the study drug
* Participant has a preplanned surgery or procedure(s) that would interfere with the conduct of the study
* Participant has received any prior treatment for IS
* Participant has been previously treated with adrenocorticotropic hormone (ACTH), corticosteroids, or Vigabatrin for seizures;
* Participant has been previously treated with a course of corticosteroids for an indication other than seizures within 30 days prior to Screening
* Participant has a known or suspected allergy to ACTH or Vigabatrin or any component of AMZ002 or Vigabatrin
* Participant has used any other investigational drug within 30 days or 5 half-lives prior to the first dose of AMZ002 or Vigabatrin (whichever is longer)
* Participant' s parent/guardian is unable to provide written informed consent and/or to complete the daily diary
* Participant has any other disease, condition, or therapy that, in the opinion of the Investigator, might compromise safety or compliance, preclude the participant from successfully completing the study, or interfere with the interpretation of the results

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Absence of Clinical Spasms as Assessed by Video Electroencephalogram (EEG) at Day 14 | At Day 14
Proportion of Participants with Resolution of Hypsarrhythmia or Significant Abnormality Compatible with Infantile Spasms (IS) as Assessed by Video EEG at Day 14 | At Day 14

SECONDARY OUTCOMES:
Time from Treatment Initiation to Absence of Clinical Spasms as Assessed by Parent/Guardian Diary | Baseline up to Day 58
Proportion of Participants with Absence of Clinical Spasms as Assessed by Parent/Guardian Diary at Day 14 | At Day 14
Proportion of Participants with Recurrence of Clinical Spasms After Initial Response as Assessed by Video EEG/ by Parent/Guardian Diary | From Day 14 up to Day 58
Time from Initial Response to Recurrence of Clinical Spasms | From Day 14 up to Day 58

CONTACTS AND LOCATIONS:
Locations (41):
- United States (12):
  - The Childrens Hospital Colorado, Aurora, Colorado
  - Miami Children's Hospital, Miami, Florida
  - Advent Health Orlando, Orlando, Florida
  - Arnold Palmer Hospital For Children, Orlando, Florida
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Kentucky Hospital, Lexington, Kentucky
  - Children's Brain Institute, Lexington, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Staten Island University Hospital, North, Staten Island, New York
  - Wake Forest Baptist Medical Center - PPDS, Winston-Salem, North Carolina
  - UT Southwestern Medical Center, Dallas, Texas
- Argentina (3):
  - Fundacion para la Lucha contra las Enfermedades Neurologicas de la Infancia, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Paediatric Hospital Dr. Juan P. Garrahan, Buenos Aires
- France (5):
  - CHU Bordeaux - Hopital des Enfants, Bordeaux
  - HFME-Hospices Civils de Lyon, Bron
  - Hopital Roger Salengro - CHU de Lille, Lille
  - Hopital Necker - Enfants Malades, Paris
  - Hopital de Hautepierre, Strasbourg
- India (4):
  - All India Institute of Medical Sciences, New Delhi, Dehli
  - Indira Gandhi Institute of Child Health, Bangalore, Karnataka
  - Amrita Advanced Centre for Epilepsy, Kochi, Kerala
  - Bharati Vidyapeeth Deemed University - Bharati Hospital, Pune, Maharashtra
- Italy (9):
  - Azienda Ospedaliero Universitaria, Ancona
  - Pediatric Hospital G. Salesi, Ancona
  - AOU Anna Meyer - Clinica di Neurologia Pediatrica, Florence
  - Istituto Pediatrico Giannina Gaslini, Genova
  - Ospedale dei Bambini Vittore Buzzi, Milan
  - Universita degli Studi di Napoli Federico II, Naples
  - Ospedale Pediatrico Bambino Gesu, Roma
  - Policlinico Universitario A.Gemelli, Roma
  - Azienda Ospedaliera Universitaria Integrata, Verona
- Mexico (3):
  - Neurociencias Estudios Clinicos S.C., Culiacán
  - HSRT, Mexico City
  - Tecnologico De Monterrey - Hospital Zambrano Hellion - Instituto de Neurologia y Neurocirugia, Nuevo León
- Poland (4):
  - The University Clinical Center, Gdansk, Gdansk
  - Provincial Specialist Children's Hospital st. Ludwika, Krakow, Krakow
  - Medical University of Warsaw, Warsaw
  - Institute of Mother and Child, Warsaw
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain